CLINICAL TRIAL: NCT07148661
Title: A Novel Technique to Remove Iatrogenic Pulmonary Parenchymal Chest Tube (PPcT): A Retrospective Analysis From a Tertiary Care Thoracic Surgery Centre
Acronym: PPcT
Status: Completed | Type: Observational
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Zeeshan Sarwar, Principal Investigator, University of Health Sciences Lahore
Other Study IDs: IRB/2025/1654/SIMS
Record Dates: First submitted 2025-08-23; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Iatrogenic Injury; Iatrogenic Disease
Keywords: Pulmonary Parenchymal chest Tube PPcT; Lung Parenchymal Injury; hemodynamic Instability; Removal of Chest Tube; Video Assisted Thoracoscopic Surgery (VATS); Thoracotomy
MeSH Terms: conditions — Iatrogenic Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PPcT Group: Participants that have been diagnosed with Iatrogenic injury to lung in case of Pulmonary Parenchymal chest tube (PPcT)
  Interventions: Procedure: Removal of PPcT

INTERVENTIONS:
Procedure: Removal of PPcT — Iatrogenic Pulmonary Parenchymal Chest Tube is removed as a staged procedure in which gradual retraction of 2cm of chest tube is done from lung parenchyma keeping an eye on the hemodynamic status of Patient.

SUMMARY:
Iatrogenic Pulmonary Parenchymal chest Tube (PPcT) placement is a recognized but underreported complication of tube thoracostomy, described both in the subcontinent and worldwide. This complication occurs when the chest tube inadvertently traverses the pleural cavity and penetrates the lung parenchyma. Patients with underlying lung pathology are at increased risk of having iatrogenic pulmonary parenchymal chest tube. In this study we describe the safe and minimally invasive technique to remove the PPcT without the need of video assisted thoracic surgery (VATS) or thoracotomy.

DETAILED DESCRIPTION:
Patients with reduced pulmonary compliance, underlying lung consolidation, or dense pleural adhesions are particularly vulnerable because these conditions limit the normal displacement of the lung away from the chest wall, predisposing it to injury during tube placement.

Diagnosing PPcT is often challenging because the clinical presentation and radiographic findings are nonspecific, and the condition may be overlooked, particularly in patients with pre-existing pulmonary disease. Computed tomography (CT) of the chest remains the gold standard for accurate diagnosis.

At our institution, we have developed and successfully implemented a stepwise, minimally invasive technique for the safe removal of PPcT over the last 19 years (since 2006), thereby avoiding thoracotomy or other invasive procedures. Once PPcT is confirmed by CT scan-while carefully differentiating true parenchymal tube placement from tubes merely located within fissures-we adopt a three-stage removal strategy:

Initial healing phase: The tube is left in situ for approximately two weeks to allow for local fibrosis and healing around the injured parenchyma, which reduces the risk of bleeding and air leak during subsequent manipulation.

Gradual staged retraction: After this period, the tube is retracted by approximately 2 cm and secured again. In cases where the tube is tightly adherent, it is rotated 360° along its axis to release any fibrous adhesions. The patient is then observed for 24 hours, with close monitoring for hemodynamic instability, hemorrhage, or air leak, and a chest radiograph is obtained to confirm tube position.

Subsequent retractions: If the patient remains stable, they are discharged and readmitted at 7-day intervals for further staged retractions of approximately 2 cm each. This process continues until the fenestrations ("eyes") of the tube exit the pleural cavity, at which point the tube is safely removed. In many cases, the tube can be removed after the first or second stage if the fenestrations have already cleared the pleural space, thereby preventing pneumothorax.

This technique has consistently yielded excellent results in our experience, allowing safe removal of PPcT while minimizing morbidity and eliminating the need for thoracotomy or video-assisted thoracoscopic surgery (VATS) for tube retrieval.

ELIGIBILITY:
Inclusion Criteria:

* All Participants having PPcT diagnosed on radiological basis is included in this study.

Exclusion Criteria:

* Participnts having normally placed pleural chest tubes. Participants having chest tubes placed in fissures of the lung diagnosed on CT Scan of chest.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with PPcT after chest tube thoracostomy either admitted to the thoracic surgery ward, emergency department, outpatient department and referred to Thoracic surgery department during the study period will be included.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Hemodynamic Instability | 24 hours
  Hemodynamic Instability after staged removal of chest tube is defined as pulse rate of greater than 120/min, systolic Blood pressure of less than 80 mm of Hg, respiratory rate of greater than 24/min, hemorrhage and persistent air leak in the chest tube. Participants were observed for these above mentioned changes after every staged retraction of chest tube and responses recorded. For the participants who develop hemodynamic instability, thoracotomy was performed and underlying cause for hemodynamic instability is addressed.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Shoaib Nabi, Clinical Professor, Principal Investigator — Services Institute of Medical Sciences (SIMS), Services Hospital, Lahore
Locations (1):
- Services Institute of Medical Sciences(SIMS), Services Hospital., Lahore, Punjab Province, Pakistan